CLINICAL TRIAL: NCT04430530
Title: 4SCAR-T Therapy After Anti-CD19 Immunotherapy Targeting B Cell Acute Lymphoblastic Leukemia
Brief Title: 4SCAR-T Therapy Post CD19-targeted Immunotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: ShiJiaZhuang Zhongxi Children Hospital (Unknown); Shenzhen Children's Hospital (Other Government); The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20008
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: CD19 Negative B-cell Malignancies
Keywords: 4S CAR-T CD22; 4S CAR-T CD123; 4S CAR-T CD38; 4S CAR-T CD10; 4S CAR-T CD20; CD19 Negative B cell leukemiaB-ALL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR-CD22/CD123/CD38/CD10/CD20 infusion (Experimental): Patients who have relapsed after anti-CD19 immunotherapy or have CD19 negative B cell malignancies
  Interventions: Biological: Infusion of 4SCAR-T specific to CD22/CD123/CD38/ CD10/CD20

INTERVENTIONS:
Biological: Infusion of 4SCAR-T specific to CD22/CD123/CD38/ CD10/CD20 — Patients who have relapsed after anti-CD19 immunotherapy or have CD19 negative B cell malignancies

SUMMARY:
This study will evaluate safety and efficacy of a combination of 4th generation chimeric antigen receptor gene-modified T cells (4SCAR-T) targeting CD19-negative B-ALL that express alternative surface antigens such as CD22, CD10, CD20, CD38, and CD123, as many patients relapse after anti-CD19 immunotherapy. Clinical response and optiminzation of a standardized lentiviral vector and cell production protocol will be investigated. This is a phase I/II trial enrolling patients from multiple clinical centers.

DETAILED DESCRIPTION:
Anti-CD19 immunotherapy based on antibody conjugated drugs or CD19-CAR-T cells has demonstrated unprecedented positive response in relapsing/refractory B-cell acute lymphoblastic leukemia (r/r B-ALL). However, many patients still relapse and up to 30-50% of those relapses are characterized by the loss of CD19 surface antigen. Patients with CD19-negative relapse usually have a poor prognosis. The mechanisms underlying CD19-negative relapses are not fully understood and it is important to develop solutions to supplement post-CD19 immunotherapies.

Potential markers for recurrent leukemic blasts in an emerging CD19-negative blast population include many known B-cell lineage antigens. To prevent further target escape and improve the therapeutic effects, the 4th generation CAR gene-modified T cells targeting CD22, CD10, CD20, CD38, or CD123 have been considered in post anti-CD19 treatment. This study aims to evaluate safety and efficacy of administrating one or multiple non-CD19 targeting CAR-T cells to patients with CD19-escaped B cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. B cell malignancies relapsed after anti-CD19 immunotherapy.
3. Malignant B cells expressing one or more of the following surface molecules: CD22/CD123/CD38/CD10/CD20.
4. The KPS score over 80 points, and survival time is more than 1 month.
5. Greater than Hgb 80 g/L.
6. No contraindications to blood cell collection.

Exclusion Criteria:

1. Complications with other active diseases, and difficult to assess patient response.
2. Bacterial, fungal, or viral infection unable to control.
3. Living with HIV.
4. Active HBV and HCV infection.
5. Pregnant and nursing mothers.
6. Under systemic steroid use within a week of the treatment.
7. Judged difficult to cooporate for continued evaluation.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of fourth generation anti-CD22/CD123/CD38/CD10/CD20 CAR-T cells | 24 weeks
  Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Anti-tumor activity of fourth generation anti-CD22/CD123/CD38/CD10/CD20 CAR-T cells | 1 year
  Scale of CAR copies are detected by qPCR and leukemic cell burden are assessed by flow cytometry

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - The Seventh Affilliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong
  - Shijiazhuang Zhongxi Children Hospital, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No